CLINICAL TRIAL: NCT06532825
Title: Cardiac Autonomic Dysfunction As a Sign of Irreversible Advanced Heart Failure
Acronym: CADYSH
Status: Recruiting | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Helena DOMINGUEZ, MD, PhD, Consultant, Assoc.Prof., University Hospital Bispebjerg and Frederiksberg
Other Study IDs: H-24002374
Record Dates: First submitted 2024-07-22; First posted 2024-08-01 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure
Keywords: heart failure; decompensated
MeSH Terms: conditions — Heart Failure | interventions — Heart Rate Determination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: heart monitoring — individual comparison of heart rate variability at admission with a repeated measurement before discharge
  Other Names: heart rate variability

SUMMARY:
The main hypothesis is that autonomic dysfunction cannot improve among patients reaching end-stage heart failure. To evaluate this, patients admitted with acute decompensated heart failure in Bispebjerg hospital, and history one or more admissions with the same condition within the prior year, will undergo repeated brief heart monitoring (10 min). Baseline recordings (at admission) will be compared with equivalent measurements before discharge to explore whether heart rate variability increases. Patients will be followed for six months after discharge from the hospital.

DETAILED DESCRIPTION:
If the patient accepts to participate and signed the project informed consent, their clinical record will be followed until the last patient included has been followed for six months.

ELIGIBILITY:
Inclusion Criteria:

* 18-years age or older
* admitted with acute decompensated heart failure for less than 48 h

Exclusion Criteria:

* pacemaker
* not signed informed consent
* other heart rhythm than sinus rhythm or atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the hospital with acute decompensated heart failure, regardless of measured left ventricle ejection fraction.
  Patients will be grouped according to rhythm: sinus rhythm and atrial fibrillation.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
number of rehospitalizations | up to six months after discharge from index admission
  number of emergency rehospitalizations, classified according to:
  1. new decompensation of heart failure
  2. side effects / complications to therapy for heart failure
  3. other

SECONDARY OUTCOMES:
Heart rate Variability change from admission to discharge | repeated measurement at baseline (within 48h from time of index admission) and before discharge (estimated one week on average from index admission)
  Measurement of heart-rate oscillations over a short term (30 min) of continuous three-lead electrocardiogram recording divided into two time domains:
  Domain 10min: relaxed, supine position for 10 min Domain 30 min: comprising the first 10 min-domain in addition to stand-up and walking for 5 min, followed by sitting relaxed until completing 30 min recording in total

OTHER OUTCOMES:
Diastolic function | six months
  Measurement of changes diastolic function in right and left ventricle based on wavelet-ECG measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology department Y, Bispebjerg-Frederiksberg Hospital, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided